CLINICAL TRIAL: NCT00293371
Title: A Phase I/II Study of Docetaxel/Prednisone and PTK 787/ZK 222584 in Previously Untreated Metastatic Hormone Refractory Prostate Cancer
Brief Title: Docetaxel, Prednisone, and Vatalanib in Treating Patients With Advanced Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456195; UCSF-04557
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Prednisone; vatalanib

INTERVENTIONS:
Drug: docetaxel
Drug: prednisone
Drug: vatalanib

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vatalanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving vatalanib together with docetaxel and prednisone may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of vatalanib when given together with docetaxel and prednisone and to see how well they work in treating patients with advanced prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicities and maximum tolerated dose of vatalanib when used in combination with docetaxel and prednisone in patients with chemotherapy-naive, metastatic, hormone-refractory prostate cancer. (phase I)

Secondary

* Determine alterations in pharmacokinetics of docetaxel and vatalanib in these patients. (phase I)
* Determine the clinical efficacy of this regimen as measured by declines in prostate-specific antigen, measurable disease response, time to progression, and overall survival. (phase II)

OUTLINE: This is a phase I open-label, dose-escalation study of vatalanib* followed by a phase II study.

* Phase I: Patients receive docetaxel IV over 1 hour on day 2. Patients also receive oral prednisone twice daily and oral vatalanib once daily on days 1-21. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
* Cohorts of 3-6 patients receive escalating doses of vatalanib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

NOTE: *Vatalanib is administered on days 5-21 during the first course only.

* Phase II: Patients receive prednisone, docetaxel, and vatalanib at the MTD as in phase I. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 93 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented adenocarcinoma of the prostate
* Progressive, systemic (metastatic) disease despite castrate levels of testosterone due to orchiectomy or luteinizing-hormone releasing hormone (LHRH) agonist, meeting 1 of the following criteria:

  * Measurable disease, defined as any lesion that can be accurately measured in at least 1 dimension ≥ 2 cm by conventional techniques or ≥ 1 cm by spiral CT scan or MRI
  * Nonmeasurable disease with PSA ≥ 5 ng/mL

    * Bone lesions
    * Pleural or pericardial effusions, ascites
    * CNS lesions, leptomeningeal disease
    * Irradiated lesions, unless progression documented after radiotherapy
    * No PSA ≥ 5 ng/mL as only evidence of disease
  * PSA evidence for progressive prostate cancer consists of a PSA level ≥ 5 ng/mL that has risen on ≥ 2 successive occasions, ≥ 2 weeks apart
* Castrate levels of testosterone (< 50 ng/dL) must be maintained

  * If no prior orchiectomy, patients must remain on testicular androgen suppression (e.g., with an LHRH analogue)
* Patients receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression after discontinuation of antiandrogen

  * Disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values, obtained at least 2 weeks apart, or documented osseous or soft tissue progression

    * For patients receiving flutamide or megestrol acetate, at least 1 of the PSA values must be obtained 4 weeks or more after flutamide/megestrol acetate discontinuation
    * For patients receiving bicalutamide or nilutamide, at least 1 of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation
  * If improvement after antiandrogen withdrawal is noted, disease progression must be established
* No pleural effusion or ascites that causes respiratory compromise ( ≥ grade 2 dyspnea)
* No history of CNS disease, including primary brain tumor, seizures, or carcinomatous meningitis

PATIENT CHARACTERISTICS:

* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* Karnofsky performance status ≥ 60%
* Life expectancy > 12 weeks
* Granulocyte count > 1,500/mm^3
* Platelet count > 75,000/mm^3
* Hemoglobin > 8.0 g/dL
* Creatinine < 1.5 times upper limit of normal (ULN)
* Bilirubin < 1.5 times ULN
* SGOT/SGPT < 1.5 times ULN
* Urinalysis ≤ 1+ proteinuria based on dipstick reading OR 2+ proteinuria on dipstick reading AND total urinary protein ≤ 3,500 mg on 24 hour urine collection and creatinine clearance ≥ 50 mL/min on a 24-hour urine collection
* No impairment of gastrointestinal (GI) function or GI disease that may affect or alter absorption of vatalanib (i.e., malabsorption syndromes)
* No myocardial infarction or significant change in anginal pattern within the last 6 months, symptomatic congestive heart failure (New York Heart Association class III or IV), or uncontrolled cardiac arrhythmia
* No pre-existing grade 3 or 4 clinical peripheral neuropathy
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No deep vein thrombosis or pulmonary embolus within the past year
* No poorly controlled diabetes (fasting blood glucose > 250) despite optimization of medical therapy
* No labile or poorly controlled hypertension (systolic blood pressure > 160 mm Hg, diastolic blood pressure > 90 mm Hg) despite maximal management with anti-hypertensives
* No serious uncontrolled, concurrent medical illness, including ongoing or active infection

  * Patients on Suppressive antibiotic therapy for chronic urinary tract infection are eligible
* No psychiatric illness or social situation that would limit compliance with treatment
* No "currently active" second malignancy other than nonmelanoma skin cancers

  * Not considered "currently active" if competed therapy and at < 30% risk of relapse
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No grapefruit or grapefruit juice during study treatment
* No history of gastrectomy/small bowel resection
* At least 4 weeks since prior hormonal therapy, including ketoconazole, aminoglutethimide, systemic steroids (any dose), and megestrol acetate (any dose)
* At least 4 weeks since prior drug or herbal product known to decrease PSA levels (e.g., finasteride, saw palmetto, or PC-SPES)
* At least 4 weeks since prior major surgery and fully recovered
* At least 4 weeks since prior radiation therapy and fully recovered
* At least 8 weeks since the last dose of prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium
* Patients receiving bisphosphonate therapy prior to initiating protocol treatment must have received bisphosphonates for at least the past month

  * No bisphosphonate initiation for 1 month prior to and during study treatment
* No prior systemic chemotherapy for prostate cancer
* No prior antiangiogenic agents (thalidomide, bevacizumab)
* No other concurrent chemotherapy, investigational agents, radiotherapy (including palliative), or biologic therapy
* No biologic therapy or immunotherapy ≤ 4 weeks prior to study treatment
* No more than 1 prior therapy with an investigational agent, completed ≥ 4 weeks prior to study treatment
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent therapeutic warfarin or similar oral anticoagulant that is metabolized by the cytochrome p450 system

  * Heparin is allowed
* No other concurrent hormonal therapy except for the following:

  * Steroids for adrenal failure
  * Hormones for nondisease-related conditions (e.g., insulin for diabetes)
  * Intermittent dexamethasone

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2005-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Time to prostate-specific antigen (PSA) and objective progression
Response rate (PSA and objective)
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Eric J. Small, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Comprehensive Cancer Center, San Francisco, California, United States